CLINICAL TRIAL: NCT00768989
Title: A Multicenter, Randomized, Open-Label, Active-Controlled Pilot Study to Evaluate the Safety and Antiretroviral Activity of Unboosted Atazanavir BID Plus Raltegravir BID and Boosted Atazanavir QD in Combination With Tenofovir/Emtricitabine QD in Treatment Naive HIV-Infected Subjects
Brief Title: Phase IIB Pilot of Atazanavir + Raltegravir
Acronym: SPARTAN
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Efficacy endpoint met, but overall experimental dosing regimen not considered optimal to support further clinical development in this population.
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI424-376
Record Dates: First submitted 2008-10-06; First posted 2008-10-08 (Estimated); Results first posted 2012-01-16 (Estimated); Last update posted 2012-02-24 (Estimated); Status verified 2012-02

CONDITIONS: HIV
Keywords: Combination Therapy
MeSH Terms: interventions — Atazanavir Sulfate; Raltegravir Potassium; Ritonavir; Tenofovir; Emtricitabine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atazanavir + Raltegravir (Experimental): Atazanavir 300 mg twice daily + Raltegravir 400 mg twice daily
  Interventions: Drug: Atazanavir; Drug: Raltegravir
- Atazanavir + Ritonavir + Tenofovir /Emtricitabine (Active Comparator): Atazanavir, 300 mg once daily, + Ritonavir, 100 mg once daily, + Tenofovir 300 mg/Emtricitabine, 200 mg once daily
  Interventions: Drug: Atazanavir; Drug: Ritonavir; Drug: Tenofovir/Emtricitabine

INTERVENTIONS:
Drug: Atazanavir — Capsules, Oral, 300 mg, twice daily, 96 weeks
  Other Names: Reyataz; BMS-232632
  Arms: Atazanavir + Raltegravir
Drug: Raltegravir — Tablet, Oral, 400 mg, twice daily, 96 weeks
  Arms: Atazanavir + Raltegravir
Drug: Atazanavir — Capsules, Oral, 300 mg, once daily, 96 weeks
  Other Names: Reyataz; BMS-232632
  Arms: Atazanavir + Ritonavir + Tenofovir /Emtricitabine
Drug: Ritonavir — Capsules, Oral, 100 mg, once daily, 96 weeks
  Arms: Atazanavir + Ritonavir + Tenofovir /Emtricitabine
Drug: Tenofovir/Emtricitabine — Tablet, Oral, 300-mg Tenofovir/200-mg Emtricitabine, once daily, 96 weeks
  Other Names: Truvada
  Arms: Atazanavir + Ritonavir + Tenofovir /Emtricitabine

SUMMARY:
The purpose of this study is to determine if the combination of atazanavir and raltegravir taken together is safe and effective in the treatment of human immunodeficiency virus (HIV).

ELIGIBILITY:
Inclusion Criteria:

* Human Immunodeficiency Virus (HIV)-1 positive status
* HIV ribonucleic acid (RNA) level >=5000 copies/mL
* Antiretroviral treatment-naive
* Absolute Cluster of Differentiation 4 (CD4) cell count meeting 1 of the following criteria:
* <350 cells/mm^3
* Screening CD4 >=350 and <=500 cells/mm^3 ONLY if at least 1 of the following conditions apply:

  * Screening HIV RNA level >100,000 copies/mL, or
  * CD4 decline >50-100 cells/mm^3/year, or
  * Age >=55 years
* Any CD4 cell count, if participant has a history of an acquired immune deficiency syndrome-defining illness
* Medically stable

Exclusion Criteria:

* Screening HIV genotype showing resistance to any component of the study regimen (Atazanavir, Raltegravir, Tenofovir/Emtricitabine)
* Hepatitis B or hepatitis C coinfection
* History of or current cardiac disease
* Electrocardiogram findings:
* PR Interval >260 msec (severe 1st degree atrioventricular block)
* QRS Interval >120 msec

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2008-11; Primary Completion 2010-01 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (15):
- United States (9):
  - Southwest Center For HIV/AIDS, Phoenix, Arizona
  - Yale University School Of Medicine, New Haven, Connecticut
  - Dupont Circle Physicians Group, Washington D.C., District of Columbia
  - Orlando Immunology Center, Orlando, Florida
  - The Aaron Diamond AIDS Research Center, New York, New York
  - University Of Cincinnati, Cincinnati, Ohio
  - Tarrant County Infectious Disease Associates, Fort Worth, Texas
  - Therapeutic Concepts, P.A., Houston, Texas
  - Diversified Medical Practices, P.A., Houston, Texas
- Argentina (4):
  - Local Institution, Buenos Aires, Bs As, Buenos Aires
  - Local Institution, Capital Federal, Buenos Aires
  - Local Institution, Mar del Plata, Buenos Aires
  - Local Institution, Rosario, Santa Fe Province
- France (2):
  - Local Institution, Nantes
  - Local Institution, Paris

REFERENCES:
- [Derived] Kozal MJ, Lupo S, DeJesus E, Molina JM, McDonald C, Raffi F, Benetucci J, Mancini M, Yang R, Wirtz V, Percival L, Zhang J, Zhu L, Arikan D, Farajallah A, Nguyen BY, Leavitt R, McGrath D, Lataillade M, The Spartan Study Team. A nucleoside- and ritonavir-sparing regimen containing atazanavir plus raltegravir in antiretroviral treatment-naive HIV-infected patients: SPARTAN study results. HIV Clin Trials. 2012 May-Jun;13(3):119-30. doi: 10.1310/hct1303-119. PMID 22592092
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from sites in Argentina (n=21 randomized), France (n=26 randomized), and the United States (n=47 randomized).
Pre-assignment Details: Of 167 participants enrolled, 94 were randomized to treatment; 1 withdrew consent after randomization but prior to study dosing. Of the 73 not randomized, 5 withdrew consent, 1 lost to follow up; 1 poor/noncompliance; 61 no longer met study criteria, and 5 for other reasons. The trial was terminated early.
Groups:
- Atazanavir + Raltegravir: Atazanavir 300 mg twice daily plus Raltegravir 400 mg twice daily
- Atazanavir + Ritonavir + Tenofovir/Emtricitabine: Atazanavir, 300 mg once daily, plus Ritonavir, 100 mg once daily, plus fixed-dose Tenofovir/emtricitabine, 300 mg/200 mg once daily
Period: Prior to Week 24
Arm/Group | Atazanavir + Raltegravir | Atazanavir + Ritonavir + Tenofovir/Emtricitabine
Started | 63 | 30
Completed | 59 | 27
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 3 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 0 | 2
Period: Week 24 to Prior to Week 36
Arm/Group | Atazanavir + Raltegravir | Atazanavir + Ritonavir + Tenofovir/Emtricitabine
Started | 59 | 27
Completed | 51 | 27
Not Completed | 8 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 6 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: On or After Week 36
Arm/Group | Atazanavir + Raltegravir | Atazanavir + Ritonavir + Tenofovir/Emtricitabine
Started | 51 | 27
Completed | 0 | 0
Not Completed | 51 | 27
Not completed — Lack of Efficacy | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Poor Compliance | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Did not attend termination visit | 2 | 0
Not completed — Sponsor Termination | 45 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atazanavir + Raltegravir | Atazanavir + Ritonavir + Tenofovir/Emtricitabine | Total
Number analyzed (Participants) | 63 | 30 | 93
Age Continuous [Mean (Standard Deviation); unit: years] | 39.5 (10.90) | 41.6 (10.87) | 40.2 (10.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 2 | 10
  Male | 55 | 28 | 83
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 6 | 14
  White | 54 | 23 | 77
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
HIV RNA Level at Baseline [Mean (Standard Deviation); unit: log10 copies/mL] | 4.9 (0.57) | 4.9 (0.66) | 4.9 (0.60)
HIV RNA Distribution at Baseline [Number; unit: Participants]
  < 30,000 copies/mL | 14 | 7 | 21
  30,000 to <100,000 copies/mL | 15 | 10 | 25
  100,000 to <500,000 copies/mL | 26 | 10 | 36
  >=500,000 copies/mL | 8 | 3 | 11
Mean Cluster of Differentiation 4 (CD4) Cell Count at Baseline [Mean (Standard Deviation); unit: cells/mm^3] | 256.2 (116.79) | 261.2 (134.93) | 257.8 (122.21)
CD4 Distribution at Baseline [Number; unit: Participants]
  < 50 cells/mm^3 | 5 | 4 | 9
  50 to < 100 cells/mm^3 | 1 | 1 | 2
  100 to < 200 cells/mm^3 | 13 | 3 | 16
  200 to < 350 cells/mm^3 | 29 | 13 | 42
  350 to < 500 cells/mm^3 | 14 | 9 | 23
  >= 500 cells/mm^3 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Human Immunodeficiency Virus (HIV) Ribonucleic Acid (RNA) Level <50 Copies/mL at Week 24
Description: The number of HIV 1-infected treatment-naive participants with an HIV RNA level <50 copies/mL after 24 weeks of treatment. Confirmed virologic response noncompleter=failure (NC=F); noncompleter=missing (NC=M); virologic response-observed cases (VR-OC).
Time Frame: At Week 24 from Baseline
Population: All randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Groups:
- Atazanavir + Raltegravir: Atazanavir, 300 mg twice daily, plus Raltegravir, 400 mg twice daily
Arm/Group | Atazanavir + Raltegravir | Atazanavir + Ritonavir + Tenofovir/Emtricitabine
Number analyzed (Participants) | 63 | 30
Participants
  NC=F (n=63, 30) | 47 | 19
  NC=M (n=58, 27) | 47 | 19
  VR-OC (n=52, 25) | 41 | 19

2. Secondary Outcome: Number of Nonresponders at Week 8
Description: Participants were classified as nonresponders if they had an HIV RNA level ≥400 copies/mL and a decrease from baseline <2 log10 copies/mL.
Time Frame: At Week 8 from Baseline
Population: The first 60 participants randomized, who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Atazanavir + Raltegravir | Atazanavir + Ritonavir + Tenofovir/Emtricitabine
Number analyzed (Participants) | 37 | 20
Participants | 0 | 1

3. Secondary Outcome: Number of Participants With HIV RNA Levels <50 Copies/mL at Weeks 48 and 96
Description: Participant HIV RNA level was determined at Weeks 48 and 96 using the Roche Amplicor® Ultrasensitive Assay Version 1. VR-OC=Virologic response-observed cases.
Time Frame: At Weeks 48 and 96 from Baseline
Population: The study terminated early, and this analysis was done only at Week 48 using VR-OC for participants who reached Week 48 when the study was terminated.
Measure: Number; unit: Participants
Groups:
- Atazanavir + Raltegravir: Atazanavir, 300 mg twice daily, plus Raltegravir 400 mg twice daily
Arm/Group | Atazanavir + Raltegravir | Atazanavir + Ritonavir + Tenofovir/Emtricitabine
Number analyzed (Participants) | 45 | 25
Participants | 37 | 19

4. Secondary Outcome: Number of Participants With HIV RNA Levels <400 Copies/mL at Week 24
Description: NC=F: noncompleter=failure; NC=M: noncompleter=missing; VR-OC: virologic response-observed
Time Frame: At Week 24 from Baseline
Population: All randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Atazanavir + Raltegravir | Atazanavir + Ritonavir + Tenofovir/Emtricitabine
Number analyzed (Participants) | 63 | 30
Participants
  NC=F (n= 63, 30) | 52 | 26
  NC=M (n=58, 27) | 52 | 26
  VR-OC (n=52, 25) | 46 | 24

5. Secondary Outcome: Number of Participants With HIV RNA Levels <400 Copies/mL at Week 48
Time Frame: At Week 48 from Baseline
Population: The study terminated early, and this analysis was only done at Week 48 using VR-OC for participants who reached Week 48 when the study was terminated.
Measure: Number; unit: Participants
Arm/Group | Atazanavir + Raltegravir | Atazanavir + Ritonavir + Tenofovir/Emtricitabine
Number analyzed (Participants) | 45 | 25
Participants | 45 | 25

6. Secondary Outcome: Number of Participants With HIV RNA Levels <400 Copies/mL at Week 96
Time Frame: At Week 96 from Baseline
Population: This analysis was not preformed due to early termination of the study.
Measure: Number; unit: Participants
Arm/Group | Atazanavir + Raltegravir | Atazanavir + Ritonavir + Tenofovir/Emtricitabine
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Mean Change From Baseline in Absolute Cluster of Differentiation 4 Cell Count
Time Frame: From Baseline to Weeks 2, 4, 8, 12, 16, 20, and 24
Population: All randomized participants who received at least 1 dose of study medication and had baseline and timepoint results.
Measure: Mean (Standard Error); unit: cells/mm^3
Arm/Group | Atazanavir + Raltegravir | Atazanavir + Ritonavir + Tenofovir/Emtricitabine
Number analyzed (Participants) | 63 | 30
cells/mm^3
  Mean change from Baseline at Week 2 (n=59, 26) | 81.1 (11.886) | 63.1 (14.248)
  Mean change from Baseline at Week 4 (n=62, 27) | 82.7 (12.238) | 100.1 (19.481)
  Mean change from Baseline at Week 8 (n=60, 29) | 111.5 (12.297) | 111.9 (16.845)
  Mean change from Baseline at Week 12 (n=62, 28) | 128.6 (13.964) | 129.3 (20.460)
  Mean change from Baseline at Week 16 (n=58, 27) | 143.6 (12.789) | 127.6 (19.336)
  Mean change from Baseline at Week 20 (n=58, 24) | 166.5 (12.189) | 140.7 (19.919)
  Mean change from Baseline at Week 24 (n=55, 24) | 166.0 (16.954) | 127.0 (17.788)

8. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Death as Outcome, AEs Leading to Discontinuation, SAEs Leading to Discontinuation
Description: AE=any new untoward medical occurrence or worsening of a preexisting medical condition that does not necessarily have a causal relationship with this treatment. SAE=any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, results in drug dependency or drug abuse, or is an important medical event.
Time Frame: Week 1 to Week 96, continuously
Population: All randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Atazanavir + Raltegravir | Atazanavir + Ritonavir + Tenofovir/Emtricitabine
Number analyzed (Participants) | 63 | 30
Participants
  AEs | 60 | 29
  SAEs | 7 | 2
  Deaths | 0 | 0
  AEs leading to discontinuation | 4 | 1
  SAEs leading to discontinuation | 1 | 0

9. Secondary Outcome: Baseline and Mean Change From Baseline in Total Cholesterol Levels
Description: The mean change from baseline in participant fasting lipids was determined using fasting serum samples.
Time Frame: From Baseline to Week 24 and Week 48
Population: All randomized participants who received at least 1 dose of study medication. N=number of participants analyzed; n=number of participants with measurements for that time point.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Atazanavir + Raltegravir | Atazanavir + Ritonavir + Tenofovir/Emtricitabine
Number analyzed (Participants) | 63 | 30
mg/dL
  Baseline (n=56, 26) | 164.6 (3.833) | 169.6 (6.756)
  Mean change from Baseline at Week 24 (n=51, 20) | 14.7 (4.367) | 15.1 (6.827)
  Mean change from Baseline at Week 48 (n=38, 20) | 18.0 (3.040) | 17.1 (4.526)

10. Secondary Outcome: Mean Change From Baseline in Total Bilirubin Level
Time Frame: From Baseline to Week 24 and Week 48
Population: All randomized participants who received at least 1 dose of study medication.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Atazanavir + Raltegravir | Atazanavir + Ritonavir + Tenofovir/Emtricitabine
Number analyzed (Participants) | 63 | 30
mg/dL
  Mean change from Baseline at Week 24 | 2.15 (0.2032) | 1.71 (0.2234)
  Mean change from Baseline at Week 48 | 2.08 (0.2176) | 1.52 (0.2206)

11. Secondary Outcome: Mean Change From Baseline in Electrocardiogram Findings
Description: The incidence of QRS wave widening and QT and PR prolongation on participant electrocardiogram findings were evaluated at study Week 24.
Time Frame: From Baseline to Week 24
Population: All randomized participants who received at least 1 dose of study medication.
Measure: Mean (Standard Error); unit: msec
Arm/Group | Atazanavir + Raltegravir | Atazanavir + Ritonavir + Tenofovir/Emtricitabine
Number analyzed (Participants) | 63 | 30
msec
  QRS Interval | 8.9 (1.019) | 3.6 (1.966)
  QTc Friderica Interval | -2.7 (2.001) | 6.0 (3.760)
  PR Interval | 17.6 (2.101) | 4.9 (2.248)

12. Secondary Outcome: Atazanavir Maximum Observed Plasma Concentration (Cmax) in 1 Dosing Interval
Description: Serial blood samples were collected over a 12-hour period after the morning dose at Week 2.
Time Frame: At Week 2 from Baseline
Population: All randomized participants who received at least 1 dose of study medication and were evaluable.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Atazanavir + Raltegravir
Number analyzed (Participants) | 13
ng/mL | 3506.5 (1366)

13. Secondary Outcome: Raltegravir Cmax in 1 Dosing Interval
Description: Serial blood samples were collected over a 12-hour period after the morning dose at Week 2.
Time Frame: At Week 2 from Baseline
Population: All randomized participants who received at least 1 dose of study medication and were evaluable.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Atazanavir + Raltegravir
Number analyzed (Participants) | 13
ng/mL | 1577.0 (2516)

14. Secondary Outcome: Atazanavir Time of Maximum Observed Plasma Concentration (Tmax)
Description: Serial blood samples were collected over a 12-hour period after the morning dose at Week 2.
Time Frame: At Week 2 from Baseline
Population: All randomized participants who received at least 1 dose of study medication and who were evaluable.
Measure: Geometric Mean (Full Range); unit: Hours
Arm/Group | Atazanavir + Raltegravir
Number analyzed (Participants) | 13
Hours | 3.0 [2.0 to 4.0]

15. Secondary Outcome: Raltegravir Tmax
Description: Serial blood samples were collected over a 12-hour period after the morning dose at Week 2.
Time Frame: At Week 2 from Baseline
Population: All randomized participants who received at least 1 dose of study medication and who were evaluable.
Measure: Geometric Mean (Full Range); unit: Hours
Arm/Group | Atazanavir + Raltegravir
Number analyzed (Participants) | 13
Hours | 2.08 [0.0 to 8.0]

16. Secondary Outcome: Atazanavir Trough Plasma Concentration (Cmin) 12 Hours Postdose
Time Frame: At Week 2 from Baseline
Population: All randomized participants who received at least 1 dose of study medication and who were evaluable.
Measure: Geometric Mean (Standard Deviation); unit: ng•h/mL
Arm/Group | Atazanavir + Raltegravir
Number analyzed (Participants) | 13
ng•h/mL | 687.1 (402)

17. Secondary Outcome: Raltegravir Cmin 12 Hours Postdose
Time Frame: At Week 2 from Baseline
Population: All randomized participants who received at least 1 dose of study medication and who were evaluable.
Measure: Geometric Mean (Standard Deviation); unit: ng•h/mL
Arm/Group | Atazanavir + Raltegravir
Number analyzed (Participants) | 13
ng•h/mL | 76.2 (94.5)

18. Secondary Outcome: Atazanavir Cmin Prior to the Morning Dose
Time Frame: At Week 2 from Baseline
Population: All randomized participants who received at least 1 dose of study medication and who were evaluable.
Measure: Geometric Mean (Standard Deviation); unit: ng*h / mL
Arm/Group | Atazanavir + Raltegravir
Number analyzed (Participants) | 13
ng*h / mL | 879.25 (495)

19. Secondary Outcome: Raltegravir Cmin Prior to the Morning Dose
Time Frame: At Week 2 from Baseline
Population: All randomized participants who received at least 1 dose of study medication and who were evaluable.
Measure: Geometric Mean (Standard Deviation); unit: ng•h/mL
Arm/Group | Atazanavir + Raltegravir
Number analyzed (Participants) | 13
ng•h/mL | 445.42 (577)

20. Secondary Outcome: Atazanavir Area Under the Concentration Curve From Time 0 to 12 Hours (AUC [0-12h]) in 1 Dosing Interval
Time Frame: At Week 2 from Baseline
Population: All randomized participants who received at least 1 dose of study medication and who were evaluable.
Measure: Geometric Mean (Standard Deviation); unit: ng•h/mL
Arm/Group | Atazanavir + Raltegravir
Number analyzed (Participants) | 13
ng•h/mL | 19903.4 (8088)

21. Secondary Outcome: Raltegravir AUC (0-12h) in 1 Dosing Interval
Time Frame: At Week 2 from Baseline
Population: All randomized participants who received at least 1 dose of study medication and who were evaluable.
Measure: Geometric Mean (Standard Deviation); unit: ng•h/mL
Arm/Group | Atazanavir + Raltegravir
Number analyzed (Participants) | 13
ng•h/mL | 6446.4 (6432)

22. Secondary Outcome: Atazanavir Area Under the Concentration Curve From Time 0 to 24 Hours (AUC [0-24h]) in 1 Dosing Interval
Description: AUC (0-24h) was estimated by multiplying AUC (0-12h) by 2.
Time Frame: At Week 2 from Baseline
Population: All randomized participants who received at least 1 dose of study medication and who were evaluable.
Measure: Geometric Mean (Standard Deviation); unit: ng•h/mL
Arm/Group | Atazanavir + Raltegravir
Number analyzed (Participants) | 13
ng•h/mL | 39806.7 (16176)

23. Secondary Outcome: Atazanavir Individual Inhibitory Quotient (IQ)
Description: Individual IQ was defined at Cmin at Week 2 divided by the protein binding adjusted EC90 (ie, the drug concentration observed to inhibit virion production by 90% in a cell-based assay) values for Atazanavir that were derived from individual participant clinical isolates.
Time Frame: At Week 2 from Baseline
Population: All randomized participants who received at least 1 dose of study medication and who were evaluable.
Measure: Geometric Mean (Full Range); unit: Units on a Scale
Arm/Group | Atazanavir + Raltegravir
Number analyzed (Participants) | 12
Units on a Scale | 23.47 [12.0 to 50.1]

24. Secondary Outcome: Atazanavir Terminal Elimination Half Life
Time Frame: At Week 2 from Baseline
Population: All randomized participants who received at least 1 dose of study medication and who were evaluable.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Atazanavir + Raltegravir
Number analyzed (Participants) | 13
Hours | 5.0 (2.2)

25. Secondary Outcome: Raltegravir Terminal Elimination Half Life
Time Frame: At Week 2 from Baseline
Population: All randomized participants who received at least 1 dose of study medication and who were evaluable.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Atazanavir + Raltegravir
Number analyzed (Participants) | 13
Hours | 2.9 (2.8)

26. Secondary Outcome: Number of Participants With Hematology Laboratory Test Results With Worst Toxicity of Grades 1 to 4 Among All Treated Participants
Description: ULN=upper limit of normal. Hematocrit(%) Grade (Gr) 1: ≥28.5-<31; Gr 2: ≥24-<28.5; Gr 3: ≥19.5-<24; Gr 4: <19.5. Hemoglobin (g/dL) Gr 1: 9.5-11; Gr 2: 8-9.4; Gr 3: 6.5-7.9; Gr 4: <6.5. Platelets (/mm^3) Gr 1: 75,000-99,000; Gr 2: 50,000-74,999; Gr 3: 20,000-49,999; Gr 4: <20,000. White Blood Cells (/mm^3) Gr 1: >2500-4000; Gr 2: >1000-<2500; Gr 3: >800-<1000; Gr 4: <800. . Prothrombin time (seconds) Gr 1: 1.01-1.25*ULN; Gr 2: 1.26-1.5*ULN; Gr 3: 1.51-3*ULN; Gr 4: >3*ULN.
Time Frame: While on treatment from Baseline through Week 96
Population: All randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Atazanavir + Raltegravir | Atazanavir + Ritonavir + Tenofovir/Emtricitabine
Number analyzed (Participants) | 63 | 30
Participants
  Hematocrit | 1 | 0
  Hemoglobin | 2 | 0
  Platelets | 1 | 1
  Prothrombin Time | 12 | 7
  White Blood Cells | 22 | 14

27. Secondary Outcome: Number of Participants With Blood Chemistry Laboratory Test Results With Worst Toxicity of Grades 1 to 4
Description: Blood urea nitrogen Gr 1:1.25-2.5*ULN;Gr 2:2.6-5.0*ULN; Gr 3:5.1-10*ULN; Gr 4:>10*ULN. Creatinine (mg/dL) Gr 1: 1.1-1.5 *ULN; Gr 2: 1.6-3*ULN: Gr 3: 3.1-6*ULN; Gr 4: >6*ULN. Hypercarbia (meq/L)Gr 1: 33-36; Gr 2:37-40; Gr 3: 41-45; Gr 4:>45. Hypocarbia (meq/L)Gr 1:19-21; Gr 2: 15-18; Gr 3: 10-14; Gr 4:<10. Hypercalcemia (mg/dL)Gr 1:10.6-11.5;Gr 2:11.6-12.5; Gr 3:12.6-13.5;Gr 4: >13.5. Hypocalcemia (mg/dL)Gr 1: 8.4-7.8;Gr 2:7.7-7; Gr 3:6.9-6.1; Gr 4: <6.1.Hyperchloremia(meq/L)Gr 1:113-116; Gr 2:117-120; Gr 3:121-125; Gr 4: >125.Hypochloremia(meq/L)Gr 1: 90-93; Gr 2: 85-89; Gr 3:80-84; Gr 4:<80.
Time Frame: While on treatment from Baseline through Week 96
Population: All randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Atazanavir + Raltegravir | Atazanavir + Ritonavir + Tenofovir/Emtricitabine
Number analyzed (Participants) | 63 | 30
Participants
  Blood urea nitrogen | 0 | 1
  Creatinine | 3 | 2
  Hypercarbia | 1 | 1
  Hypocarbia | 15 | 7
  Hypercalcemia | 2 | 1
  Hypocalcemia | 1 | 1
  Hyperchloremia | 0 | 0
  Hypochloremia | 1 | 1
  Hyperkalemia | 2 | 0
  Hypokalemia | 6 | 5
  Hypernatremia | 0 | 0
  Hyponatremia | 3 | 1
  Hyperclycemia | 8 | 5
  Hypoglycemia | 6 | 4

28. Secondary Outcome: Number of Participants With Blood Chemistry Laboratory Test Results With Worst Toxicity of Grades 1 to 4 (Continued)
Description: Hyperkalemia(meq/L) Gr 1: 5.6-6; Gr 2: 6.1-6.5; Gr 3: 6.6-7; Gr4: >7. Hypokalemia(meq/L) Gr 1: 3-3.4; Gr 2: 2.5-2.9; Gr 3: 2-2.4; Gr 4:<2. Hypernatremia (meq/L) Gr 1: 148-150; Gr 2: 151-157; Gr 3: 148-165; Gr 4: >165. Hyponatremia (meq/L) Gr 1: 130-132; Gr 2: 123-129; Gr 3: 116-122; Gr 4: >115.Hyperglycemia(mg/dL)Gr 1: 116-160; Gr 2: 161-250; Gr 3: 251-500; Gr 4: >500. Hypoglycemia(mg/dL)Gr 1: 55-64; Gr 2: 40-54; Gr 3:30-39;Gr 4:<30.Creatine kinase (IU/L) Gr 1: >ULN-1.5*ULN; Gr 2: 1.5-3*ULN; Gr 3: >3-6*ULN; Gr 4: >6.0*ULN. Albumin (g/dL) Gr 1: <LLN-30; Gr 2: <30-20; Gr 3&4: <20.
Time Frame: While on treatment from Baseline through Week 96
Population: All randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Atazanavir + Raltegravir | Atazanavir + Ritonavir + Tenofovir/Emtricitabine
Number analyzed (Participants) | 63 | 30
Participants
  Hyperkalemia | 2 | 1
  Hypokalemia | 1 | 1
  Hypernatremia | 0 | 0
  Hyponatremia | 3 | 1
  Hyperclycemia | 8 | 5
  Hypoglycemia | 6 | 4
  Creatine kinase | 21 | 7
  Albumin | 3 | 2

29. Secondary Outcome: Number of Participants With Enzyme and Urine Laboratory Test Results With Worst Toxicity of Grades 1 to 4
Description: AST/SGOT=Aspartate aminotransferase/serum glutamate oxaloacetate transaminase; ALT/SGPT=Alanine transaminase/serum glutamic pyruvic transaminase. Bilirubin (mg/dL)Gr 1: 1.1-1.5*ULN;Gr 2:1.6-2.5*ULN;Gr3:2.6-5*ULN;Gr4:>5*ULN.AST/SGOT(U/L)Gr 1:1.25-2.5*ULN;Gr 2: 2.6-5*ULN;Gr 3:5.1-10*ULN;Gr4:>10*ULN.ALT/SGPT (U/L)Gr 1:1.25-2.5*ULN;Gr 2:1.4-2.09*ULN;Gr 3:5.1-10*ULN;Gr4:>10*ULN. Lipase(U/L)Gr 1:1.1-1.39*ULN;Gr 2:>1.5-2*ULN;Gr 3:2.5-5;Gr 4:5*ULN.Proteinuria(g/24 hr loss)Gr 1:1+or <1;Gr 2:2-3+or>1-2; Gr 3:4+or>2-3.5;Gr4:>3.5.Creatine kinase(IU/L)Gr1:2-3*ULN;Gr 2:3.1-5*ULN;Gr 3:5.1-10*ULN;Gr4:>10*ULN.
Time Frame: While on treatment from Baseline through Week 96
Population: All randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Atazanavir + Raltegravir | Atazanavir + Ritonavir + Tenofovir/Emtricitabine
Number analyzed (Participants) | 63 | 30
Participants
  Total Bilirubin | 62 | 28
  AST/SGOT | 11 | 8
  ALT/ SGPT | 10 | 8
  Lipase | 11 | 13
  Proteinurea | 14 | 11
  Creatine kinase | 21 | 7

ADVERSE EVENTS:
Time Frame: While on treatment from Baseline through Week 96
Arm/Group | Atazanavir + Ritonavir + Tenofovir/Emtricitabine | Atazanavir + Raltegravir
Serious Adverse Events (participants affected / at risk) | 7/63 | 2/30
Other Adverse Events (participants affected / at risk) | 58/63 | 27/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atazanavir + Ritonavir + Tenofovir/Emtricitabine (N=63) | Atazanavir + Raltegravir (N=30)
B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BURNS FIRST DEGREE (Injury, poisoning and procedural complications) | 1 | 0
ATRIAL FLUTTER (Cardiac disorders) | 1 | 0
KAPOSI'S SARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
MALARIA (Infections and infestations) | 0 | 1
OVERDOSE (Injury, poisoning and procedural complications) | 1 | 0
SUICIDE ATTEMPT (Psychiatric disorders) | 1 | 0
TESTIS CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
DEPRESSION (Psychiatric disorders) | 1 | 0
GUN SHOT WOUND (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Atazanavir + Ritonavir + Tenofovir/Emtricitabine (N=63) | Atazanavir + Raltegravir (N=30)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 | 2
OCULAR ICTERUS (Eye disorders) | 15 | 4
ABDOMINAL PAIN (Gastrointestinal disorders) | 4 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 | 5
ASTHENIA (General disorders) | 2 | 2
BRONCHITIS (Infections and infestations) | 9 | 3
FATIGUE (General disorders) | 4 | 5
HAEMORRHOIDS (Gastrointestinal disorders) | 5 | 0
HERPES ZOSTER (Infections and infestations) | 4 | 2
TOOTH INFECTION (Infections and infestations) | 4 | 2
BILIRUBIN CONJUGATED INCREASED (Investigations) | 10 | 2
BLOOD BILIRUBIN INCREASED (Investigations) | 11 | 3
NASOPHARYNGITIS (Infections and infestations) | 4 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 3 | 2
SINUSITIS (Infections and infestations) | 5 | 0
VOMITING (Gastrointestinal disorders) | 3 | 2
ACARODERMATITIS (Infections and infestations) | 0 | 2
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 6 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 | 3
DIARRHOEA (Gastrointestinal disorders) | 8 | 5
HEADACHE (Nervous system disorders) | 11 | 3
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 2
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 4 | 1
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 8 | 4
INSOMNIA (Psychiatric disorders) | 1 | 3
NAUSEA (Gastrointestinal disorders) | 3 | 7
PARAESTHESIA (Nervous system disorders) | 1 | 2
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 3
PRURITUS (Skin and subcutaneous tissue disorders) | 4 | 3
COUGH (Respiratory, thoracic and mediastinal disorders) | 6 | 8
INFLUENZA (Infections and infestations) | 2 | 4
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 2
SYPHILIS (Infections and infestations) | 4 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 6 | 6
CONJUNCTIVITIS (Eye disorders) | 0 | 2
FLATULENCE (Gastrointestinal disorders) | 1 | 2
GENITAL HERPES (Infections and infestations) | 4 | 1
JAUNDICE (Hepatobiliary disorders) | 15 | 2
PYREXIA (General disorders) | 4 | 1
RASH (Skin and subcutaneous tissue disorders) | 8 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication